CLINICAL TRIAL: NCT04638647
Title: An Open-label, Multi-center Protocol for Patients Who Have Completed a Previous Novartis Sponsored Secukinumab Study and Are Judged by the Investigator to Benefit From Continued Secukinumab Treatment
Brief Title: Secukinumab Open Label Roll-over Extension Protocol
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAIN457A02001B; 2023-504417-67-00 (Registry Identifier: EU CT NUMBER)
Record Dates: First submitted 2020-11-16; First posted 2020-11-20 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Autoimmunity, Inflammation
Keywords: Secukinumab, Post trial access
MeSH Terms: conditions — Autoimmune Diseases; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Secukinumab s.c. (Experimental): Participants will be started on 75 mg, 150 mg or 300 mg s.c. Q4W depending on what dose the participant was receiving in the parent trial (for trials with i.v. formulation the starting dose will be 300 mg s.c.). The study medication dose may be modified basedu pon clinical need, the judgement of the investigator and health authority guidelines (if applicable). For pediatric participants, the dose should not be increased beyond the maximum dose evaluated in the respective weight category in the parent protocol.
  Interventions: Biological: Secukinumab s.c. injection

INTERVENTIONS:
Biological: Secukinumab s.c. injection — Secukinumab pre-filled syringes (PFS) for s.c. injection

SUMMARY:
The purpose of this study is to assess long term safety in participants who have completed a Novartis trial with secukinumab, have been judged by the investigator to benefit from continued treatment with secukinumab, and are unable to obtain the marketed secukinumab formulation.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent must be obtained for adult participants before any assessment is performed. Written informed assent and parental permission (age as per local law) must be obtained for pediatric participants before any assessment is performed. If participants reach age of consent (age as per local law) during the study, they will need to also sign the corresponding study informed consent(s).
2. Ability to communicate effectively with the investigator, to understand and willing to comply with the requirements of the study.
3. Participant has completed treatment per protocol in a Novartis study of secukinumab (unless otherwise specified in a parent study protocol). Participants, who derive benefit from the treatment with secukinumab but have not completed the treatment in certain parent studies, due to parent study termination by Novartis, may be eligible if the termination was due to reasons other than safety or lack of efficacy (technical / administrative reasons).
4. Participant is deriving benefit from secukinumab, investigator believes he/she would continue to derive benefit from secukinumab and the benefit outweighs the risk, based on the investigator's judgement.
5. Participant is unable to obtain access to the marketed secukinumab formulation per local prescription and/or reimbursement guidelines.

Exclusion Criteria:

1. Participant has prematurely discontinued study treatment in the parent protocol.
2. Women of childbearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using methods of contraception during the entire study or longer if required by locally approved prescribing information (e.g., in European Union (EU) 20 weeks).

Ages: 6 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2020-12-22 (Actual); Primary Completion 2030-01-29 (Estimated); Study Completion 2030-04-04 (Estimated)

PRIMARY OUTCOMES:
To evaluate long term safety as assessed by occurrence of AEs/SAEs | up to 2 years
  Serious adverse events (SAEs), adverse events (AEs), and injection site reactions

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (132):
- United States (28):
  - Providence Medical Foundation, Fullerton, California
  - Purushotham Akther and Roshan Kotha MD Inc, La Mesa, California
  - Precn Comprehensive Clnl Rsch Solns, San Leandro, California
  - Orrin Troum MD and Medical Associates, Santa Monica, California
  - Inland Rheumatology Clinical Trials INC, Upland, California
  - Medvin Clinical Research, Van Nuys, California
  - Center for Rheumatology Research, West Hills, California
  - Denver Arthritis Clinic, Denver, Colorado
  - Rheumatology Associates of South Florida, Boca Raton, Florida
  - Homestead Assoc In Research Inc, Homestead, Florida
  - IRIS Research and Development, Plantation, Florida
  - Conquest Research, Winter Park, Florida
  - FL Medical Clinic Orlando Health, Zephyrhills, Florida
  - Willow Rheumatology Wellness, Willowbrook, Illinois
  - Dawes Fretzin Clinical Rea Group, Indianapolis, Indiana
  - Klein and Associates, Hagerstown, Maryland
  - Ahmed Arif Medical Research Center, Grand Blanc, Michigan
  - Physician Research Collaboration, Lincoln, Nebraska
  - Arthritis Rheumatology and Bone Disease Associates PA, Voorhees Township, New Jersey
  - St Lawrence Health System, Potsdam, New York
  - Oregon Health Sciences University, Portland, Oregon
  - Altoona Center for Clin Res, Duncansville, Pennsylvania
  - West Tennessee Research Institute, Jackson, Tennessee
  - Austin Regional Clinic Rheumatology, Austin, Texas
  - Southwest Rheum Rsrch LLC, Mesquite, Texas
  - Accurate Clinical Research Inc, San Antonio, Texas
  - Overlake Arthritis and Osteoporosis, Bellevue, Washington
  - Rheumatology Pulmonary Clinic, Beckley, West Virginia
- Brazil (6):
  - Novartis Investigative Site, Vitória, Espírito Santo
  - Novartis Investigative Site, Salvador, Estado de Bahia
  - Novartis Investigative Site, Juiz de Fora, Minas Gerais
  - Novartis Investigative Site, São Paulo, São Paulo
  - Novartis Investigative Site, Rio de Janeiro
  - Novartis Investigative Site, Sao Jose Rio Preto
- Bulgaria (4):
  - Novartis Investigative Site, Pleven
  - Novartis Investigative Site, Plovdiv
  - Novartis Investigative Site, Sofia
  - Novartis Investigative Site, Stara Zagora
- China (28):
  - Novartis Investigative Site, Hefei, Anhui
  - Novartis Investigative Site, Beijing, Beijing Municipality
  - Novartis Investigative Site, Chongqing, Chongqing Municipality
  - Novartis Investigative Site, Xiamen, Fujian
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Shantou, Guangdong
  - Novartis Investigative Site, Shenzhen, Guangdong
  - Novartis Investigative Site, Wuhan, Hubei
  - Novartis Investigative Site, Changsha, Hunan
  - Novartis Investigative Site, Zhuzhou, Hunan
  - Novartis Investigative Site, Baotou, Inner Mongolia
  - Novartis Investigative Site, Hohhot, Inner Mongolia
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Yangzhou, Jiangsu
  - Novartis Investigative Site, Nanchang, Jiangxi
  - Novartis Investigative Site, Pingxiang, Jiangxi
  - Novartis Investigative Site, Changchun, Jilin
  - Novartis Investigative Site, Linyi, Shandong
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Ürümqi, Xinjiang
  - Novartis Investigative Site, Kunming, Yunnan
  - Novartis Investigative Site, Ningbo, Zhejiang
  - Novartis Investigative Site, Wenzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Bengbu
  - Novartis Investigative Site, Jinan
  - Novartis Investigative Site, Shanghai
  - Novartis Investigative Site, Tianjin
- Colombia (4):
  - Novartis Investigative Site, Bogota, Cundinamarca
  - Novartis Investigative Site, Chía, Cundinamarca
  - Novartis Investigative Site, Bucaramanga, Santander Department
  - Novartis Investigative Site, Ibagué, Tolima Department
- Czechia (7):
  - Novartis Investigative Site, Ostrava, Czech Republic
  - Novartis Investigative Site, Brno-Zidonice, CZE
  - Novartis Investigative Site, Prague, Prague 1
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Hradec Králové
  - Novartis Investigative Site, Prague
  - Novartis Investigative Site, Uherské Hradiště
- Novartis Investigative Site, Pátrai, Greece
- Novartis Investigative Site, Guatemala City, Guatemala
- India (6):
  - Novartis Investigative Site, Surat, Gujarat
  - Novartis Investigative Site, Bangalore, Karnataka
  - Novartis Investigative Site, Mumbai, Maharashtra
  - Novartis Investigative Site, Nashik, Maharashtra
  - Novartis Investigative Site, Hyderabad, Telangana
  - Novartis Investigative Site, New Delhi
- Italy (2):
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Reggio Emilia, RE
- Malaysia (2):
  - Novartis Investigative Site, Kuching, Sarawak
  - Novartis Investigative Site, Kuala Lumpur
- Mexico (3):
  - Novartis Investigative Site, Guadalajara, Jalisco
  - Novartis Investigative Site, Culiacan, State of Mexico
  - Novartis Investigative Site, Metepec, State of Mexico
- Poland (10):
  - Novartis Investigative Site, Krakow, Lesser Poland Voivodeship
  - Novartis Investigative Site, Wroclaw, Lower Silesian Voivodeship
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Bydgoszcz
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Poznan
  - Novartis Investigative Site, Sochaczew
  - Novartis Investigative Site, Torun
  - Novartis Investigative Site, Warsaw
  - Novartis Investigative Site, Wroclaw
- Novartis Investigative Site, Lisbon, Portugal
- Russia (12):
  - Novartis Investigative Site, Barnaul
  - Novartis Investigative Site, Chelyabinsk
  - Novartis Investigative Site, Kazan'
  - Novartis Investigative Site, Kemerovo
  - Novartis Investigative Site, Krasnodar
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Saratov
  - Novartis Investigative Site, Smolensk
  - Novartis Investigative Site, Ulyanovsk
  - Novartis Investigative Site, Yaroslavl
  - Novartis Investigative Site, Yekaterinburg
- South Africa (2):
  - Novartis Investigative Site, Panorama, Western Cape
  - Novartis Investigative Site, Stellenbosch, Western Cape
- South Korea (2):
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul
- Spain (10):
  - Novartis Investigative Site, Santiago Compostela, A Coruna
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Barcelona
  - Novartis Investigative Site, Bilbao, Bizkaia
  - Novartis Investigative Site, Santander, Cantabria
  - Novartis Investigative Site, Vigo, Pontevedra
  - Novartis Investigative Site, A Coruña
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Seville
  - Novartis Investigative Site, Valencia
- Switzerland (3):
  - Novartis Investigative Site, Basel
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Sankt Gallen

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing access to patient-level data and supporting clinical documents from eligible studies with qualified external researchers. Requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to protect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com